CLINICAL TRIAL: NCT04143581
Title: Evaluating the Short-Term Renal and Systemic Effects of SGLT2 Inhibition in Non-Diabetic Patients at Risk of Accelerated GFR Decline Because of Glomerular Hyperfiltration: a Sequential OFF-ON-OFF Study With One-Month Empagliflozin Therapy Followed by One-Month Recovery Period
Brief Title: SGLT2 Inhibitors in Glomerular Hyperfiltration
Acronym: EMPATHY
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMPATHY; 2019-004152-10 (EudraCT Number)
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Non-diabetic Chronic Kidney Disease
Keywords: GFR decline; Glomerular hyperfiltration; SGLT2 inhibitors; Residual proteinuria; Obesity
MeSH Terms: conditions — Obesity | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: OFF/ON/OFF design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMP (Experimental)
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin 10 mg/die for 28 days
  Other Names: Jardiance

SUMMARY:
Glomerular hyperfiltration is a major risk factor for accelerated glomerular filtration rate (GFR) decline and renal and cardiovascular events despite optimized conservative therapy with blood pressure and blood glucose (in diabetics) lowering medications and inhibitors of the Renin Angiotensin System (RAS) such as Angiotensin Converting Enzyme (ACE) inhibitors and/or Angiotensin Receptor Blockers (ARBs).

Progressive GFR decline initiated and sustained by glomerular hyperfiltration in subjects with diabetes, unhealthy obesity, hypertension and other risk factors, is paralleled by progressive glomerulosclerosis and loss of functioning nephrons.

The inhibition of the sodium-glucose cotransporter 2 (SGLT2) in the proximal tubular segments of the nephrons appears to be an ideal, specific intervention to inhibit the tubulo-glomerular feedback and ameliorate glomerular hyperfiltration in subjects with absolute or relative hyperfiltration associated with unhealthy obesity or proteinuric chronic kidney disease (CKD). Indeed, by reducing tubular sodium reabsorption, SGLT2 inhibitors may enhance sodium chloride delivery to the macula densa, restore pre-glomerular resistances and therefore limit glomerular hyperperfusion and consequent hyperfiltration. Moreover, because of its natriuretic effects, SGLT2 inhibition therapy might reduce the sodium overload and volume expansion which, along with secondary hypertension, may further contribute to kidney hyperperfusion and glomerular hyperfiltration in obesity and CKD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years old;
2. Increased risk of accelerated renal function loss because of absolute or relative hyperfiltration associated with unhealthy obesity or residual proteinuria defined as:

   Unhealthy obesity:
   * BMI >30 kg/m^2 or waist circumference >94 cm in males and > 80 cm in females
   * Metabolic syndrome, defined as the presence of at least three of the following criteria:
   * Blood pressure>140/90 mmHg or controlled blood pressure under current antihypertensive treatment
   * Triglyceride levels >150 mg/dL
   * HDL<40 mg/dL in males <50 mg/dL in females
   * Fasting blood glucose > 100 and <125 mg/dL

   Residual proteinuria:
   * Urinary protein excretion >1g/24-h to <3g/24-h despite RAS inhibitor therapy with ACE inhibitors or ARBs;
   * Blood pressure in recommended targets with or without blood pressure lowering medications;
3. Estimated GFR > 60 ml/min/1.73m^2 (CKD-EPI formula);
4. Female childbearing potential and non-sterile male must agree to use a method of contraception;
5. Written informed consent

Exclusion Criteria:

1. Type 1or 2 diabetic patients;
2. Concomitant treatment with insulin or oral hypoglycemic agents;
3. Nephrotic syndrome of any etiology;
4. Patients with Autosomal Dominant Polycystic Kidney Disease;
5. Symptomatic urinary tract lithiasis or obstruction;
6. Ischemic kidney disease (because of possible excess risk of acute kidney injury upon SGLT2 inhibition associated reduction in sodium pool and kidney perfusion pressure);
7. Rapidly progressive kidney disease defined by impairment of renal function within 2 weeks - 3 months (for the cohort of patients with residual proteinuria only) ;
8. Active systemic autoimmune diseases;
9. Treatment for glomerulopathies or systemic diseases with steroids or any other immunosuppressive agent within one year;
10. Specific contraindication to SGLT2 inhibitor therapy;
11. Heart failure with or without decreased systolic function;
12. Uncontrolled hypertension or symptomatic hypotension;
13. History of malignancy within 5 years of screening;
14. Inability to fully understand the possible risks and benefits related to study participation;
15. If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 90 days after last dose; or intending to donate ova during such time period;
16. If male, the subject intends to donate sperm while on the study this study or for 90 days after last dose;
17. Alcohol and drug abuse;
18. Participation in another interventional clinical trial within the 4 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Measured Glomerular Filtration Rate (GFR) | Changes from baseline to the end of one-month treatment period and one-month recovery period
  GFR will be measured by the iohexol plasma clearance technique

SECONDARY OUTCOMES:
24 hour urinary output | Changes from baseline to the end of one-month treatment period and one-month recovery period
  last of three consecutive collections
24 hour urinary protein excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  mean of the measurement in three consecutive 24-hour urine collection
24 hour urinary albumin excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  mean of the measurement in three consecutive 24-hour urine collection
24 hour urinary urea excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  last of three consecutive collections
24 hour urinary phosphate excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  last of three consecutive collections
24 hour urinary sodium excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  last of three consecutive collections
24 hour urinary glucose excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  last of three consecutive collections
24 hour urinary potassium excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  last of three consecutive collections
24 hour urinary uric acid excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  last of three consecutive collections
24 hour urinary creatinine excretion | Changes from baseline to the end of one-month treatment period and one-month recovery period
  last of three consecutive collections
Fractional clearance of total protein calculated by standard formulas | Changes from baseline to the end of one-month treatment period and one-month recovery period
Fractional clearance of albumin calculated by standard formulas | Changes from baseline to the end of one-month treatment period and one-month recovery period
Fractional clearance of sodium calculated by standard formulas | Changes from baseline to the end of one-month treatment period and one-month recovery period
Fractional clearance of potassium calculated by standard formulas | Changes from baseline to the end of one-month treatment period and one-month recovery period
Fractional clearance of uric acid calculated by standard formulas | Changes from baseline to the end of one-month treatment period and one-month recovery period
Fractional clearance of free water calculated by standard formulas | Changes from baseline to the end of one-month treatment period and one-month recovery period
Glucose disposal rate | Changes from baseline to the end of one-month treatment period and one-month recovery period
  Performed by hyperinsulinemic euglycemic clamp and by standard oral glucose load and HOMA index;
Glucose tolerance | Changes from baseline to the end of one-month treatment period and one-month recovery period
  Performed by hyperinsulinemic euglycemic clamp and by standard oral glucose load and HOMA index;
Office blood pressure | Changes from baseline to the end of one-month treatment period and one-month recovery period
Office heart rate | Changes from baseline to the end of one-month treatment period and one-month recovery period
24 hour (day-time and night-time) blood pressure monitoring | Changes from baseline to the end of one-month treatment period and one-month recovery period
24 hour (day-time and night-time) heart rate monitoring | Changes from baseline to the end of one-month treatment period and one-month recovery period
Pulse wave velocity | Changes from baseline to the end of one-month treatment period and one-month recovery period
  These parameters will be measured by tonometry
other marker of vascular stiffness | Changes from baseline to the end of one-month treatment period and one-month recovery period
  These parameters will be measured by tonometry
Indices of Quality of Life: questionnaire SF-36 | Changes from baseline to the end of one-month treatment period and one-month recovery period
  By submission of validate questionnaire

IPD SHARING:
Plan to Share IPD: No